CLINICAL TRIAL: NCT06641414
Title: A Global Multicenter, Double-blind, Randomized, Registrational Phase 3 Study of Lisaftoclax (APG-2575) in Combination With Azacitidine (AZA) in Patients With Newly Diagnosed Higher Risk Myelodysplastic Syndrome (HR-MDS) (GLORA-4).
Brief Title: Lisaftoclax (APG-2575) Combined With Azacytidine (AZA) in the Treatment of Patients With Higher-risk Myelodysplastic Syndrome (GLORA-4).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APG2575MG301
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Higher-risk Myelodysplastic Syndrome
Keywords: Higher-risk Myelodysplastic Syndrome; Lisaftoclax
MeSH Terms: interventions — Lisaftoclax; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lisaftoclax (APG-2575) combined with Azacitidine (Experimental)
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: Azacitidine Injection
- Placebo combined with Azacitidine (Active Comparator)
  Interventions: Drug: Azacitidine Injection; Other: Placebo

INTERVENTIONS:
Drug: Lisaftoclax (APG-2575) — QD, oral administration.
  Arms: Lisaftoclax (APG-2575) combined with Azacitidine
Drug: Azacitidine Injection — QD, hypodermic or intravenous injection.
Other: Placebo — QD, oral administration.
  Arms: Placebo combined with Azacitidine

SUMMARY:
A global multicenter, randomized, double-blind, placebo-controlled, pivotal phase III study. To evaluate overall survival (OS) of Lisaftoclax (APG-2575) combined with azacitidine (AZA) vs. placebo combined with azacitidine in newly diagnosed patients with HR-MDS.

DETAILED DESCRIPTION:
This study intends to enroll patients with HR-MDS to receive the therapy of Lisaftoclax (APG-2575) combined with azacitidine (AZA) or placebo combined with azacitidine.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed higher-risk MDS.
2. ECOG score of ≤2.
3. Expected survival ≥ 3 months.
4. Adequate organ function.
5. Female subjects of potential childbearing potential have a negative urine or serum pregnancy test before dosing. Subjects of childbearing potential as well as their partners voluntarily use contraception deemed effective by the investigator during the treatment period and for at least six months after the last dose of study drug.
6. Able to understand and voluntarily sign a written informed consent form, which must be signed prior to the performance of any trial-specified study procedures.
7. Subjects are able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. Concomitant other malignancies or prior malignancies with disease-free intervals of less than 1 year at the time of signing the informed consent.
2. Have undergone hematopoietic stem cell transplantation.
3. Uncontrolled active infection
4. Use of moderately potent inducers and moderately potent inhibitors of CYP3A4 within 14 days prior to the first dose of study drug.
5. MDS or other conditions that cannot be administered enterally.
6. Any condition that the subject is deemed to be inappropriate to participate in this study after evaluation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS） | Up to 5 years
  The primary endpoint was overall survival (OS), defined as the time from the date of randomization to the date of death of any cause.

SECONDARY OUTCOMES:
Safety evaluation based on the adverse event concurrence | Up to 5 years
  Number of treatment emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, M.D., Ph.D., Study Chair — Peking University People's Hospital; Guillermo Garcia-Manero, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- Peking University People's Hospital, Beijing, Beijing Municipality, China